CLINICAL TRIAL: NCT05379218
Title: Remote Ischemic Conditioning in Hypoxic-Ischemic Encephalopathy: A Safety and Feasibility Trial
Brief Title: RIC in HIE: A Safety and Feasibility Trial
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The Hospital for Sick Children (Other)
Responsible Party: Principal Investigator, Brian Kalish, Neonatologist, The Hospital for Sick Children
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 1000077295
Record Dates: First submitted 2021-11-25; First posted 2022-05-18 (Actual); Last update posted 2024-03-07 (Actual); Status verified 2024-03

CONDITIONS: Hypoxic-Ischemic Encephalopathy
Keywords: Hypoxic-Ischemic Encephalopathy
MeSH Terms: conditions — Hypoxia-Ischemia, Brain

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention Arm - Remote Ischemic Conditioning (Experimental): Remote Ischemic Conditioning
  Interventions: Device: Remote Ischemic Conditioning
- Control Arm - No Remote Ischemic Conditioning (No Intervention): No intervention. A blood pressure cuff will be placed on the infant's arm but will not be inflated.

INTERVENTIONS:
Device: Remote Ischemic Conditioning — Patients randomized to the RIC arm, cohorts of 4 consecutive patients will receive escalating therapy:
  A. 4 consecutive patients will undergo 4 cycles of 3 minutes ischemia, followed by 5 minutes reperfusion, on Day 1 of therapeutic hypothermia B. Observing no safety events (see below) from patients in group A, 4 consecutive patients will undergo 4 cycles of 5 minutes ischemia, followed by 5 minutes reperfusion, on Day 1 of therapeutic hypothermia.
  C. Observing no safety events from patients in group B, 4 consecutive patients will undergo 4 cycles of 5 minutes ischemia, followed by 5 minutes reperfusion, on Days 1 and 2 of therapeutic hypothermia.
  D. Observing no safety events from patients in group C, 4 consecutive patients will undergo 4 cycles of 5 minutes ischemia, followed by 5 minutes reperfusion, on Days 1, 2, and 3 of therapeutic hypothermia.
  All infants will have an extra 1ml of blood collected.
  Arms: Intervention Arm - Remote Ischemic Conditioning

SUMMARY:
Remote Ischemic Conditioning has never been studied in neonates with HIE. However, RIC has been studied in animal models of perinatal asphyxia and has shown encouraging results. In neonatal rats with HIE, RIC is associated with reduced sensory motor deficits compared to non-RIC, and repeated cycles in three consecutive days is superior to a single treatment. In piglets, four cycles of 10 minutes of bilateral hindlimb ischemia immediately after bilateral common carotid occlusion results in reduced cell death in the periventricular white matter and internal capsule. These preclinical studies support the hypothesis that RIC may be beneficial in infants with HIE.

DETAILED DESCRIPTION:
Hypoxic-ischemic encephalopathy (HIE) is a devastating condition in which newborn infants are deprived of oxygen in the peripartum period, resulting in brain injury. HIE is a leading cause of infant morbidity and mortality worldwide. Within the last 15 years, the introduction of hypothermia as a therapy for HIE has revolutionized our care of these vulnerable infants, but despite these improvements, nearly 50% of infants die or have major disability at 18 months. Therefore, there is a significant need to develop novel adjunctive therapies for HIE.

Remote ischemic conditioning (RIC) is a procedure that involves the application of brief cycles of non-lethal ischemia and reperfusion to a remote site, with the goal of protecting distant organs exposed to ischemic injury. RIC has been extensively studied in experimental models and applied clinically in adults, children, and neonates. In neonates, there have been trials exploring its potential role before cardiac surgery and necrotizing enterocolitis. Most of these studies performed up to 4 cycles of 5 minutes of ischemia in a single day and found RIC to be feasible and safe. Experimental studies suggest that RIC, acting through three inter-related mechanisms (neural, humoral, and systemic pathways) is associated with increased cerebral blood flow, decreased inflammation, and enhanced cell survival. RIC has been studied as a potential treatment in adult stroke, and while the evidence to date is inconclusive, preliminary data suggest that RIC may reduce the size and the severity of the stroke lesion, as well as improve cognitive outcomes.

RIC has been studied in animal models of perinatal asphyxia and has shown encouraging results. In neonatal rats with HIE, RIC is associated with reduced sensory motor deficits compared to non-RIC, and repeated cycles in three consecutive days is superior to a single treatment. In piglets, four cycles of 10 minutes of bilateral hindlimb ischemia immediately after bilateral common carotid occlusion results in reduced cell death in the periventricular white matter and internal capsule. These preclinical studies support the hypothesis that RIC may be beneficial in infants with HIE. In this proposal, we outline a carefully designed and conducted early phase study of RIC in neonates with HIE.

ELIGIBILITY:
Inclusion Criteria:

* Qualifying for therapeutic hypothermia according to the primary care team based on the current SickKids HIE Protocol

Exclusion Criteria:

* Gestational age <35 weeks
* Known central nervous system malformations
* Known chromosomal or genetic anomalies
* Confirmed or suspected inborn error of metabolism
* Parental decision for withdrawal of life-sustaining treatment ("comfort care"). If this decision is made after enrollment but before completion of RIC intervention, no further study-related intervention will be performed.
* Patients requiring significant hemodynamic support (two or more agents for blood pressure support, >0.05mcg/kg/min epinephrine infusion, or >0.1 mU/kg/min vasopressin) for the four hour period prior to RIC
* Patients requiring inhaled nitric oxide or fraction of inspired oxygen (FiO2) >50% for the four-hour period prior to RIC

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2022-01-17 (Actual); Primary Completion 2024-02-05 (Actual); Study Completion 2024-02-05 (Actual)

PRIMARY OUTCOMES:
RIC cycles administered as planned (Y/N) | 72 hours
  Designated RIC cycles are administered as planned (dichotomous variable)
Incidence of Treatment-Emergent Adverse Events [Safety and Tolerability] | 72 hours
  Frequency of limb ischemia, incidence of RIC interruption and rescue intervention, incidence of subcutaneous fat necrosis, incidence of acute kidney injury, mortality

SECONDARY OUTCOMES:
Number of patients with cutaneous injury | 24 hours
  New-onset of skin breakdown, bruising, ecchymosis or petechiae, within 24 hours after the end of the maneuver (comparing to the previous baseline assessment)
Number of patients with transient and persistent pain defined as a premature infant pain profile (PIPP) score >7 | 24 hours
  Pain measured by PIPP score > 7 will be considered as an episode of pain. A patient will be considered to have persistent pain if PIPP score is higher than the baseline score 6 hours after the maneuver.

OTHER OUTCOMES:
aEEG | 4 hours
  Background pattern/s (and relative duration) before (2 hours) and after (2 hours) RIC.
  Background pattern/s include classifying the tracings by lower margin of tracing in microvolts and upper margin of tracing in microvolts. Normal aEEG pattern vs continuous normal voltage, discontinuous normal voltage, burst suppression, low voltage, or flat +/- seizures.
  Normal aEEG pattern: lower margin >5 microvolts and upper margin >10 microvolts.
  Presence of sleep-wake cycles and seizures.
Biomarkers | 72 hours
  Blood collected at 72 hours will be used to measure biomarkers for brain injury: S100B, blood brain-derived neurotrophic factor, total Tau, and neuron-specific enolase as measured in nanograms per milliliter. Blood will also be bio banked for additional immune-related analysis, but will not be used for genetic analysis.
MRI including diffusion-weighted imaging and spectroscopy | 7 days
  MRI will be done between day 4 and 7 of age, as per standard of care, and scored for injury severity. MRI will be scored according to Weeke et al. criteria (Journal of Pediatrics 2018).
Number of patients with cognitive, motor, and/or language impairment at 18-24 months corrected age defined as < 85 (impairment) and <70 (severe impairment) on the Bayley Scales of Infant and Toddler Development (3rd edition) | 18-24 months
  1. Neurodevelopment: cognitive, motor, and language impairment defined as a Bayley Scales of Infant and Toddler Development (3rd edition) scores < 85 (impairment) and <70 (severe impairment).
  2. Deafness or hearing impairment.
  3. Blindness or visual impairment.
Number of patients with deafness or hearing impairment on decibel scale at 18-24 months corrected age | 18-24 months
  Deafness or hearing impairment on decibel scale
Number of patients with blindness or visual impairment on visual acuity scale at 18-24 months corrected age | 18-24 months
  Blindness or visual impairment on visual acuity scale

CONTACTS AND LOCATIONS:
Overall Officials: Brian Kalish, MD, Principal Investigator — The Hospital for Sick Children
Locations (1):
- The Hospital for Sick Children, Toronto, Ontario, Canada